CLINICAL TRIAL: NCT03942133
Title: Ultrasound-guided Continuous Adductor Canal Block for Analgesia After Total Knee Replacement: Comparison of Block at the Entrance and Middle of the Canal
Brief Title: Tow Techniques of Adductor Canal Block for Analgesia After Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Cui Xulei, Attending physician, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CXL1
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Total Knee Arthroplasty; Analgesia; Nerve Block
Keywords: adductor canal block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- entrance placement of adductor canal catheter (Experimental)
  Interventions: Procedure: ultrasound-guided short-axis placement of catheter at the entrance of the adductor canal
- middle point placement of adductor canal catheter (Experimental)
  Interventions: Procedure: ultrasound-guided long-axis placement of catheter at the middle of the adductor canal

INTERVENTIONS:
Procedure: ultrasound-guided short-axis placement of catheter at the entrance of the adductor canal — Ultrasound probe is placed at the entrance of the adductor canal in short axis ，insertion of a PAJUNK Contiplex S catheter with the tip of the catheter located at the entrance of the canal
  Arms: entrance placement of adductor canal catheter
Procedure: ultrasound-guided long-axis placement of catheter at the middle of the adductor canal — Ultrasound probe is placed at the middle of the adductor canal in long axis with the caphelad end of the probe aligned with the entrance of the canal. insertion of a PAJUNK Contiplex S catheter with the tip of the catheter located at the middle of the canal
  Arms: middle point placement of adductor canal catheter

SUMMARY:
This study compares the tow technique of continues adductor canal block for total knee replacement surgery. Half participants will receive catheterization at the entrance of the adductor canal, while the other half will receive catheterization at the middle point of the adductor canal.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years
* Knee-arthroscopy
* Written consent
* ASA I-III
* BMI 19-35

Exclusion Criteria:

* Unable to communicate with the investigators (e.g., a language barrier or a neuropsychiatric disorder).
* coagulopathy or on anticoagulant medication
* Allergic reactions toward drugs used in the trial
* History of substance abuse
* Infection at injection site
* Can not be mobilised to 5 meters of walk pre-surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-05-11 (Actual); Primary Completion 2019-12-08 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
cumulative sulfentanil consumption at 24 hours after surgery | 24 hours after surgery

SECONDARY OUTCOMES:
the strength of quadriceps femoris | 0,2,4,8,24,48 hours postoperatively
  Quadriceps strength was assessed on a 0-5 scale as per the Medical Research Council Scale quadriceps motor strength(0 = no voluntary contraction possible, 1 = muscle flicker, but no movement of limb, 2 = active movement only with gravity eliminated, 3 = movement against gravity but without resistance, 4 = movement possible against some resistance and 5 = normal motor strength against resistance)
The pain scores at rest determined by the numeric rating scale (NRS, 0-10) | at 0,2,4,8,24,48 hours postoperatively
  11-point numerical rating scale (NRS; 0, no pain; 10, maximum pain imaginable).
The pain scores on adduction of the keen determined by the numeric rating scale (NRS, 0-10) | at 0,2,4,8,24,48 hours postoperatively
  11-point numerical rating scale (NRS; 0, no pain; 10, maximum pain imaginable).
incidence of postoperative nausea and vomiting (PONV) | within 48 hours after surgery
Patient satisfaction with anesthesia | within 5th day after surgery
  Patient satisfaction with anesthesia was assessed using a 5-point scale (5, very satisfied; 4, satisfied; 3, neither satisfied nor dissatisfied; 2, dissatisfied; 1, very dissatisfied)
complications | within 3days after surgery
  Record complications including catheter dislodgment, puncture point infection, leakage,falling down,et al.
cumulative sulfentanil consumption at other time points after surgery | 2,4,8,48 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fei Y, Cui X, Chen S, Peng H, Feng B, Qian W, Lin J, Weng X, Huang Y. Continuous block at the proximal end of the adductor canal provides better analgesia compared to that at the middle of the canal after total knee arthroplasty: a randomized, double-blind, controlled trial. BMC Anesthesiol. 2020 Oct 9;20(1):260. doi: 10.1186/s12871-020-01165-w. PMID 33036554